CLINICAL TRIAL: NCT00543881
Title: Telemedical Interventional Monitoring in Heart Failure (TIM-HF)
Brief Title: Telemedical Interventional Monitoring in Heart Failure
Acronym: TIM-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Economics and Technology (Other Government)
Responsible Party: Principal Investigator, Friedrich Koehler, Senior Physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01MG531
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Heart Failure
Keywords: telemedicine; remote patient monitoring; chronic heart failure; mortality; health economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interventional group
  Interventions: Device: Remote patient monitoring (Partnership for the Heart)
- 2 (Active Comparator): Usual care group
  Interventions: Device: Usual care group

INTERVENTIONS:
Device: Remote patient monitoring (Partnership for the Heart) — Guideline-based care in heart failure (NYHA II-III) including at least 5 scheduled doctor's visits plus daily monitoring of ECG, weight, blood pressure, self-report of health status, weekly monitoring of physical fitness
  Other Names: brand name for remote patient monitoring system: Partnership for the Heart
  Arms: 1
Device: Usual care group — Guideline-based care in heart failure (NYHA II-III) including at least 5 scheduled doctor's visits
  Arms: 2

SUMMARY:
Superiority of additional Remote Patient Monitoring in patients with CHF In comparison to usual care in terms of:

* reduction of mortality rate
* reduction of hospitalizations
* increasement of patients' quality of life

DETAILED DESCRIPTION:
The clinical trial assesses 710 patients over a period of at least 15 months each (2008 until 2010); all participants will continue to receive usual care from their GP. All patients will be examined at the beginning of the study and will undergo a check-up every 3 months. 355 of the patients will be randomly allocated to receive devices for Remote Patient Monitoring which will measure various parameters on a daily basis (e.g., weight, blood pressure, heart rate). The devices are mobile and can be used at home or elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory CHF NYHA II or III
2. LVEF ≤ 35% and cardiac decompensation with hospitalization for heart failure or therapy with intravenous diuretics (.40 mg furosemide/day) within 24 months prior to enrolment or LVEF ≤ 25%, measured twice within past 6 months
3. Optimal medical treatment for CHF (b-blocker, ACE-inhibitor/ ARB, diuretics) including ICD/CRT if indicated
4. Age ≥ 18 years
5. Informed consent

Exclusion Criteria:

1. Existence of any disease (HF excluded) reducing life expectancy to less than 1 year
2. Insufficient compliance to telemonitoring or study visits
3. Impairment to use the telemonitoring equipment or appear to study visits (e.g. dementia, impaired self-determination, lacking ability to communicate)
4. Pregnancy
5. Concurrent participation in other therapy trials
6. Hospitalization for cardiac decompensation within 7 days before inclusion in trial
7. Implanted cardiac assist system
8. Unstable angina pectoris
9. Congenital heart defect
10. Primary heart valve disease
11. Hypertrophic or restrictive cardiomyopathy
12. Arrhythmogenic right ventricular cardiomyopathy
13. Acute myocarditis diagnosis ,1 year
14. Actively listed for heart transplantation
15. Planned revascularization or CRT implantation
16. Chronic renal insufficiency with creatinine .2.5 mg/dl
17. Liver cirrhosis
18. Known alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
all cause mortality

SECONDARY OUTCOMES:
comp of the combined rate of cv death and hosp. for worsening HF;days lost due to cv death or HF hosp;cv mortality;Rate of cv hosp;Rate of hosp for HF;hosp for any reason;cv hosp;hosp for HF;duration of all hosp for HF;NYHA class; SF-36; PHQ-9 score

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Koehler, MD, Principal Investigator — Charité - Universitaetsmedizin Berlin
Locations (2):
- Germany (2):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Robert-Bosch-Krankenhaus, Stuttgart

REFERENCES:
- [Background] Koehler F, Anker SD. Noninvasive home telemonitoring: the Trans-European Network-Home-Care Management System. J Am Coll Cardiol. 2006 Aug 15;48(4):850-1; author reply 851-2. doi: 10.1016/j.jacc.2006.05.033. Epub 2006 Jul 24. No abstract available. PMID 16904569
- [Background] Kohler F, Schieber M, Lucke S, Heinze P, Henke S, Matthesius G, Pferdt T, Wegertseder D, Stoll M, Anker SD. ["Partnership for the Heart"--development and testing of a new remote patient monitoring system]. Dtsch Med Wochenschr. 2007 Mar 2;132(9):458-60. doi: 10.1055/s-2007-970358. No abstract available. German. PMID 17315125
- [Background] Winkler S, Schieber M, Lucke S, Heinze P, Schweizer T, Wegertseder D, Scherf M, Nettlau H, Henke S, Braecklein M, Anker SD, Koehler F. A new telemonitoring system intended for chronic heart failure patients using mobile telephone technology--feasibility study. Int J Cardiol. 2011 Nov 17;153(1):55-8. doi: 10.1016/j.ijcard.2010.08.038. Epub 2010 Sep 18. PMID 20851481
- [Background] Anker SD, Koehler F, Abraham WT. Telemedicine and remote management of patients with heart failure. Lancet. 2011 Aug 20;378(9792):731-9. doi: 10.1016/S0140-6736(11)61229-4. PMID 21856487
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Kim SS, Koehler K, Lucke S, Honold M, Heinze P, Schweizer T, Braecklein M, Kirwan BA, Gelbrich G, Anker SD; TIM-HF Investigators. Telemedical Interventional Monitoring in Heart Failure (TIM-HF), a randomized, controlled intervention trial investigating the impact of telemedicine on mortality in ambulatory patients with heart failure: study design. Eur J Heart Fail. 2010 Dec;12(12):1354-62. doi: 10.1093/eurjhf/hfq199. PMID 21098580
- [Result] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Baumann G, Honold M, Koehler K, Gelbrich G, Kirwan BA, Anker SD; Telemedical Interventional Monitoring in Heart Failure Investigators. Impact of remote telemedical management on mortality and hospitalizations in ambulatory patients with chronic heart failure: the telemedical interventional monitoring in heart failure study. Circulation. 2011 May 3;123(17):1873-80. doi: 10.1161/CIRCULATIONAHA.111.018473. Epub 2011 Mar 28. PMID 21444883
- [Result] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, de Brouwer S, Perrin E, Baumann G, Gelbrich G, Boll H, Honold M, Koehler K, Kirwan BA, Anker SD. Telemedicine in heart failure: pre-specified and exploratory subgroup analyses from the TIM-HF trial. Int J Cardiol. 2012 Nov 29;161(3):143-50. doi: 10.1016/j.ijcard.2011.09.007. Epub 2011 Oct 8. PMID 21982700
- [Result] Prescher S, Deckwart O, Winkler S, Koehler K, Honold M, Koehler F. Telemedical care: feasibility and perception of the patients and physicians: a survey-based acceptance analysis of the Telemedical Interventional Monitoring in Heart Failure (TIM-HF) trial. Eur J Prev Cardiol. 2013 Jun;20(2 Suppl):18-24. doi: 10.1177/2047487313487483e. PMID 23702987
- [Result] Jehn M, Prescher S, Koehler K, von Haehling S, Winkler S, Deckwart O, Honold M, Sechtem U, Baumann G, Halle M, Anker SD, Koehler F. Tele-accelerometry as a novel technique for assessing functional status in patients with heart failure: feasibility, reliability and patient safety. Int J Cardiol. 2013 Oct 12;168(5):4723-8. doi: 10.1016/j.ijcard.2013.07.171. Epub 2013 Jul 25. PMID 23962782
- [Result] Prescher S, Deckwart O, Koehler K, Lucke S, Schieber M, Wellge B, Winkler S, Baumann G, Koehler F. [Will telemonitoring be adopted by patients with chronic heart failure?]. Dtsch Med Wochenschr. 2014 Apr;139(16):829-34. doi: 10.1055/s-0034-1369849. Epub 2014 Apr 10. German. PMID 24722932
- [Result] Prescher S, Schoebel C, Koehler K, Deckwart O, Wellge B, Honold M, Hartmann O, Winkler S, Koehler F. Prognostic value of serial six-minute walk tests using tele-accelerometry in patients with chronic heart failure: A pre-specified sub-study of the TIM-HF-Trial. Eur J Prev Cardiol. 2016 Oct;23(2 suppl):21-26. doi: 10.1177/2047487316671438. PMID 27892422
- [Derived] Jehn M, Halle M, Schuster T, Hanssen H, Koehler F, Schmidt-Trucksass A. Multivariable analysis of heart rate recovery after cycle ergometry in heart failure: exercise in heart failure. Heart Lung. 2011 Nov-Dec;40(6):e129-37. doi: 10.1016/j.hrtlng.2011.01.005. Epub 2011 Mar 23. PMID 21429580
- [Derived] Jehn M, Halle M, Schuster T, Hanssen H, Weis M, Koehler F, Schmidt-Trucksass A. The 6-min walk test in heart failure: is it a max or sub-maximum exercise test? Eur J Appl Physiol. 2009 Oct;107(3):317-23. doi: 10.1007/s00421-009-1128-0. Epub 2009 Jul 18. PMID 19618202